CLINICAL TRIAL: NCT05642377
Title: A Randomized, Double-Blind, Placebo Controlled, Single and Multiple Dosing, Dose-Escalation Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic/Pharmacodynamic Characteristics and Food Effect After Oral Administration of HGR4113 in Healthy Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetic/Pharmacodynamic Characteristics and Food Effect of HGR4113 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Glaceum (Industry)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HGR4113-P1-01
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- HGR4113 300 mg Single Dose (Experimental): Single oral dosing of HGR4113 300 mg
  Interventions: Drug: HGR4113
- Placebo 300 mg Single Dose (Placebo Comparator): Single oral dosing of placebo 300 mg
  Interventions: Drug: Placebo
- HGR4113 600 mg Single Dose (Experimental): Single oral dosing of HGR4113600 mg
  Interventions: Drug: HGR4113
- Placebo 600 mg Single Dose (Placebo Comparator): Single oral dosing of placebo 600 mg
  Interventions: Drug: Placebo
- HGR4113 1200 mg Single Dose (Experimental): Single oral dosing of HGR41131200 mg
  Interventions: Drug: HGR4113
- Placebo 1200 mg Single Dose (Placebo Comparator): Single oral dosing of placebo 1200 mg
  Interventions: Drug: Placebo
- HGR4113 200 mg Multiple Dose (Experimental): Multiple oral dosing of HGR4113 200 mg, twice daily
  Interventions: Drug: HGR4113
- Placebo 200 mg Multiple Dose (Placebo Comparator): Multiple oral dosing of placebo 200 mg, twice daily
  Interventions: Drug: Placebo
- HGR4113 400 mg Multiple Dose (Experimental): Multiple oral dosing of HGR4113 400 mg, twice daily
  Interventions: Drug: HGR4113
- Placebo 400 mg Multiple Dose (Placebo Comparator): Multiple oral dosing of placebo 400 mg, twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HGR4113 — Once-daily oral administration
  Arms: HGR4113 1200 mg Single Dose; HGR4113 300 mg Single Dose; HGR4113 600 mg Single Dose
Drug: Placebo — Once-daily oral administration
  Arms: Placebo 1200 mg Single Dose; Placebo 300 mg Single Dose; Placebo 600 mg Single Dose
Drug: HGR4113 — Twice-daily oral administration
  Arms: HGR4113 200 mg Multiple Dose; HGR4113 400 mg Multiple Dose
Drug: Placebo — Twice-daily oral administration
  Arms: Placebo 200 mg Multiple Dose; Placebo 400 mg Multiple Dose

SUMMARY:
1. Study Objective: The objective of this study is to evaluate the safety, tolerability, pharmacokinetic/pharmacodynamic characteristics, and food effect of HGR4113 after single and multiple oral administration in healthy subjects.
2. Study Design and Plan: This study is a randomized, double-blind, placebo controlled, single and multiple dosing, dose-escalation phase 1 clinical trial. Volunteers who have been deemed eligible based on the inclusion/exclusion criteria will be given a random number. Each subject will be assigned to one of the dose groups in a 6:2 ratio to HGR4113 (active) or placebo. Subjects will be studied in a double-blind manner and will receive the investigational product per protocol. Dose will be escalated once safety data is collected up to the last pharmacokinetic blood collection timepoint and safety and tolerability has been deemed acceptable following the review of the Safety Review Committee. Assessments including vital signs, 12-lead ECG, clinical laboratory, reproductive hormones, physical examination, and monitoring of adverse events concomitant medications will be conducted to evaluate safety and tolerability. Blood will be collected to evaluate the pharmacokinetic/pharmacodynamic characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form approved by the IRB before Screening.
2. Adult volunteers between 19 and 50 years of age at Screening.
3. Body mass index (BMI) between 18.0 and 24.9.

   ☞ BMI (kg/m^2) = body weight (kg) / (height [m])^2
4. In good health, determined by no clinically significant findings from medical history, physical examination, vital signs, 12-lead electrocardiogram, and clinical laboratory tests at Screening, or subjects who are deemed acceptable by the Investigator regardless of the test results.

Exclusion Criteria:

1. Significant history or clinical manifestation of any hepatic, kidney, neurological, immune, respiratory, endocrine, hematological, neoplastic, or cardiovascular disease, or psychiatric disorder (e.g., mood disorder, obsessive-compulsive disorder).
2. History of stomach or intestinal disorders (e.g., Chron's disease, ulcer) or surgeries - not including appendectomy, hemorrhoidectomy, or herniotomy - which may affect the safety or pharmacokinetic/pharmacodynamic evaluation of the investigational product.
3. Significant history or clinical manifestation of hypersensitivity to any drug including licorice or other drug (e.g., aspirin, antibiotics).
4. One or more of the following laboratory test results at Screening:

   * ANC < 1000
   * AST, ALT, GGT, total bilirubin > 1.5x upper limit normal
   * Fasting glucose ≥ 126 mg/dL or HbA1c ≥ 6.5% despite two retests
   * eGFR < 60 (CKD-EPI).
5. Systolic blood pressure < 90 mmHg or > 150 mmHg, or diastolic blood pressure < 60 mgHg or > 100 mmHg as determined by vital signs monitored after resting in sitting position for at least 3 minutes.
6. History of drug/chemical abuse or tested positive in urine drug screen.
7. Used or intend to use any prescription medications/products or phytotherapeutic/herbal/plant-derived preparations within 14 days prior to dosing, or any nonprescription medications/products (i.e., over-the-counter (OTC) drugs), health products, or vitamins within 7 days prior to dosing, unless deemed acceptable by the Investigator.
8. Participation in any clinical study or bioequivalence study within 6 months prior to dosing.
9. Whole blood donation within 2 months prior to dosing, plasma/platelet donation within 1 month prior to dosing, or receipt of blood products within 1 month prior to dosing.
10. Alcohol consumption > 21 units/week (1 unit = 10 g of pure alcohol) or unable to abstain from consuming alcohol 3 days prior to first dosing until the last pharmacokinetic blood sampling.
11. History of smoking within 90 days prior to dosing (however, participation is acceptable if the subject has quit at least 90 days prior to dosing) or unable to abstain from smoking 90 days prior to dosing until the last pharmacokinetic blood sampling.
12. Ingestion of grapefruit-containing foods or beverages 24 hours 3 days prior to dosing until the last pharmacokinetic blood sampling, or unable to abstain from ingesting such foods or beverages during the same period.
13. Unable to abstain from ingesting caffeine-containing foods or beverages (e.g., coffee, tea [e.g., black tea, green tea], soft drinks, coffee milk, energy drinks, sports drinks) 3 days prior to dosing until the last pharmacokinetic blood sampling.
14. Females, excluding those who have amenorrhea for at least 12 months or have been surgically sterilized (e.g., bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), who are pregnant or lactating, evidenced by a positive urine hCG pregnancy test.
15. Subject or subject's partner is unable or unwilling to use a medically acceptable means of contraception during and for 90 days following the last dosing or willing to donate sperm during the same period.

    - Acceptable contraceptive methods include:
    * Use of an intrauterine device that has been proven highly effective
    * Male or female physical contraceptive used with chemical sterilization
    * Surgical sterilization of the subject or the subject's partner (e.g., vasectomy, hysterectomy, tubal ligation, salpingectomy).
16. Subjects who, in the opinion of the Investigator, should not participate in in this study based on other reasons.
17. Subject who is confirmed as the CYP2C19 poor metabolizer (e.g., *2/*2, *2/*3, *3/*3) by exploratory genotyping test at Screening in MAD group.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability Assessment by Adverse Event Monitoring | Day 1 to 7 days after day of last administration
  Number of participants with observed adverse events
Safety and Tolerability Assessment by Number of Patients with Change in Physical Examination | Day 1 to 7 days after day of last administration
  Number of participants with clinically significant change in physical examination
Safety and Tolerability Assessment by Number of Participants with Change in Vital Signs | Day 1 to 7 days after day of last administration
  Number of participants with clinically significant change in vital signs including blood pressure, heart rate, and body temperature
Safety and Tolerability Assessment by Number of Participants with Change in Laboratory Test | Day 1 to 7 days after day of last administration
  Number of participants with clinically significant change in laboratory test assessed through hematology, blood biochemistry, urinalysis, blood coagulation, and hormone tests
Safety and Tolerability Assessment by Number of Participants with Change in 12-Lead Electrocardiogram | Day 1 to 7 days after day of last administration
  Number of participants with clinically significant change in 12-lead electrocardiogram
Safety and Tolerability Assessment by Number of Participants with Change in Semen Parameters | From Screening to 12 weeks after day of last administration
  Number of participants with clinically significant change in semen assessed through semen volume, semen pH, sperm count, sperm concentration, sperm motility, and sperm morphology
Pharmacokinetic Assessment by Maximum Plasma Concentration of HGR4113 | Hour 0 to 96
  Maximum Plasma Concentration of HGR4113 (Cmax)
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HGR4113 Over Dosing Interval | Hour 0 to 24
  Area Under the Plasma Concentration-Time Curve of HGR4113 Over Dosing Interval (AUCtau)
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HGR4113 from Time Zero to the Last Measurable Point | Hour 0 to 96
  Area Under the Plasma Concentration-Time Curve of HGR4113 from Time Zero to the Last Measurable Point (AUClast)
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HGR4113 from Time Zero to Infinity | Hour 0 to 96
  Area Under the Plasma Concentration-Time Curve of HGR4113 from Time Zero to Infinity (AUCinf)
Pharmacokinetic Assessment by Half-Life of HGR4113 | Hour 0 to 96
  Half-life of HGR4113 (T1/2)
Pharmacokinetic Assessment by Time to Maximum Observed Plasma Concentration of HGR4113 | Hour 0 to 96
  Time to Maximum Observed Plasma of HGR4113 (Tmax)
Pharmacokinetic Assessment by Oral Clearance of HGR4113 | Hour 0 to 96
  Oral Clearance of HGR4113 (CL/F)
Pharmacokinetic Assessment by Apparent Volume of Distribution of HGR4113 | Hour 0 to 96
  Volume of Distribution of HGR4113 (Vz/F)

SECONDARY OUTCOMES:
Pharmacodynamic Assessment by Change in Paraoxonase 1 Activity | Day -1 to 17
  Change in paraoxonase 1 activity
Pharmacodynamic Assessment by Change in Plasma Glucose | Day -1 to 17
  Change in plasma glucose level
Pharmacodynamic Assessment by Change in Plasma HbA1c | Day -1 to 17
  Change in plasma HbA1c level
Pharmacodynamic Assessment by Change in Plasma Insulin | Day -1 to 17
  Change in plasma insulin level
Pharmacodynamic Assessment by Change in Plasma C-peptide | Day -1 to 17
  Change in plasma c-peptide level

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Sang Yu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No